CLINICAL TRIAL: NCT06806384
Title: Effects of Cognitive-Motor Exergame Using Dividat Senso on Physical and Cognitive Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Changho Song, Professor, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2023-10-007-001
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Stroke Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ExerGame group (Experimental): Participants in the experimental group train using the Dividat Senso platform, a pressure-sensitive device equipped with 20 sensors. They engage in ExerGames designed to improve balance, coordination, and cognitive processing speed through tasks such as weight shifting, stepping accuracy, and reaction time, with difficulty levels adjusted based on performance. A waist-high parallel bar is available for support to ensure safety during the exercises. In addition to this training, participants receive 30-minute sessions of conventional physical therapy, including range-of-motion exercises, upper-limb training, and respiratory training, five days per week over a four-week period.
  Interventions: Other: ExerGame-based Stroke Rehabilitation; Other: Conventional physical therapy for stroke rehabilitation
- General balance exercise group (Active Comparator): Participants in the general balance group follow a standardized program of balance exercises aimed at improving postural control and stability. The program includes daily 30-minute sessions of weight-shifting activities, focusing on anterior-posterior and mediolateral movements, with an emphasis on loading the affected limb. Exercises involve forward-backward lunges, lateral movements with parallel foot positioning, and standing on a balance pad to enhance postural stability. In addition to the balance exercises, participants also receive conventional physical therapy, including range-of-motion exercises, upper-limb training, and respiratory training, provided for 30 minutes per day, five days per week, over four weeks.
  Interventions: Other: General balance exercise for stroke rehabilitation; Other: Conventional physical therapy for stroke rehabilitation

INTERVENTIONS:
Other: ExerGame-based Stroke Rehabilitation — The intervention involves training using the Dividat Senso platform (Dividat, Schindellegi, Switzerland), a pressure-sensitive platform (1.13 m × 1.13 m) equipped with 20 sensors. The training includes a series of ExerGames designed to challenge balance, coordination, and cognitive processing speed. These games focus on weight shifting, stepping accuracy, and reaction time, with difficulty levels progressively adjusted based on participant performance. To ensure safety, participants are allowed to use a waist-high parallel bar for support during the exercises. Additionally, participants receive conventional physical therapy methods that do not interfere with the study protocol. These include range-of-motion exercises, upper-limb training, and respiratory training, delivered in 30-minute sessions, five days per week, over a four-week period.
  Arms: ExerGame group
Other: General balance exercise for stroke rehabilitation — The intervention consists of a standardized program of balance exercises designed to improve postural control and stability. The program incorporates weight-shifting training performed once daily for 30 minutes, five days per week, over a four-week period. Weight-shifting activities include anterior-posterior and mediolateral movements, with a focus on loading the affected limb. Participants are instructed to adopt a lunge posture for forward-backward movements, maintain parallel foot positioning for lateral movements, and utilize a balance pad to enhance postural stability. A trained therapist adjusts the intensity and difficulty of the exercises to match the individual abilities of each participant, ensuring a personalized and progressive approach.
  Arms: General balance exercise group
Other: Conventional physical therapy for stroke rehabilitation — The intervention includes conventional physical therapy methods that are compatible with the study protocol. These methods consist of range-of-motion exercises, upper-limb training, and respiratory training. The sessions are delivered for 30 minutes per day, five days per week, over a four-week period.

SUMMARY:
The objective of this randomized controlled trial is to assess whether exergaming using the Dividat Senso platform more effectively enhances physical and cognitive functions in patients with chronic stroke compared to standard balance exercises. The primary questions it seeks to answer are:

* Does exergaming with the Dividat Senso lead to greater improvements in physical function, as measured by outcomes such as the Functional Gait Assessment and the Short Physical Performance Battery?
* Does exergaming with the Dividat Senso result in greater enhancements in cognitive function, evaluated through measures such as the Trail Making Test (Parts A and B) and the Stroop Test?

Researchers will compare two groups:

* An ExerGame group, receiving exergaming with the Dividat Senso in addition to standard rehabilitation.
* A Control group, receiving standard balance exercises.

Participants will:

* Undergo a four-week training period, consisting of five sessions per week, with each session lasting 30 minutes.
* Receive standard rehabilitation, including neurodevelopmental treatment and occupational therapy, alongside their assigned balance or exergame exercises.
* Complete baseline and post-intervention assessments of physical function (using the Functional Gait Assessment and the Short Physical Performance Battery) and cognitive function (using the Trail Making Test and the Stroop Test).
* During each exergame session, participants in the ExerGame group will interact with the Dividat Senso platform, performing weight-shifting, stepping, and task-oriented balancing exercises guided by real-time feedback on a virtual interface.
* Participants in the Control group will perform standard balance exercises emphasizing weight transfer in anterior-posterior and medial-lateral directions.

This study aims to clarify the efficacy of exergaming as a dual-task intervention for chronic stroke rehabilitation, potentially offering a more engaging and effective approach to improving both motor and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic stroke (≥6 months post-stroke) confirmed by medical records
* a score of 21 or higher on the Korean version of the Mini-Mental State Examination
* ability to walk independently ≥10 meters with or without assistive devices

Exclusion Criteria:

* hemianopia
* other neurological disorders (e.g., Parkinson's disease, multiple sclerosis)
* progressive or uncontrolled medical conditions (e.g., unstable cardiac disease, uncontrolled diabetes)
* musculoskeletal conditions that could interfere with balance or gait performance
* participation in other interventional studies within the past year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Functional Gait Assessment | Baseline, after four weeks
  The Functional Gait Assessment is an instrument designed to assess postural stability during ambulation and the individual's ability to perform various tasks while walking. Scores are assigned on an ordinal scale from 0 to 3, with a total score of 30.

SECONDARY OUTCOMES:
Short Physical Performance Battery | Baseline, after four weeks
  The Short Physical Performance Battery is a physical performance test used to assess lower extremity function in older adults. It consists of three components: balance, gait speed, and chair stand (5 repetitions). Each task is scored from 0 (inability to perform) to 4, based on performance differences, with a maximum total score of 12. Although this tool is commonly used to quantify lower extremity function in older adults, it can also assess more challenging endurance-based long-distance performance, differentiating it from traditional clinical assessment tools for stroke patients
Trail Making Test A and B | Baseline, after four weeks
  The Trail Making Test consists of two parts: Part A, in which participants connect 25 numbered circles on a page, and Part B, in which participants alternately connect numbered and lettered circles. Trail Making Test-A measures visual scanning and processing speed, while Trail Making Test-B assesses divided attention, set-shifting, and cognitive flexibility. The participants' reaction times (in seconds) and the number of errors were recorded.
Stroop Test | Baseline, after four weeks
  The Stroop Test assesses selective attention and interference sensitivity. It consists of three parts: a page with color names printed in matching ink colors, a page with meaningless symbols (X's) printed in various ink colors, and a page with color names printed in incongruent ink colors (e.g., the word "blue" printed in red ink). In this study, the third part (incongruent color names) was used for testing, and the participants' completion time and the number of errors were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Seoul, Nowon-gu, South Korea